CLINICAL TRIAL: NCT03023969
Title: Implication of Two Different Doses of Intradiscal O2-O3 Injection Upon the Pain Alleviation in Patients With Low Back Pain: A Randomized, Single-blind Study
Brief Title: Implication of Two Doses of O2-O3 Upon the Pain Alleviation in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00009908
Record Dates: First submitted 2017-01-12; First posted 2017-01-18 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Active Comparator): percutaneous ozone intradiscal injection group A receive 10 ml of ozone oxygen mixture 40 ug O3/ ml O2
  Interventions: Drug: ozone oxygen mixture
- group B (Active Comparator): percutaneous ozone intradiscal injection group receive 10 ml of ozone oxygen mixture 30 ug O3/ ml O2.
  Interventions: Drug: ozone oxygen mixture

INTERVENTIONS:
Drug: ozone oxygen mixture — receive 10 ml of ozone oxygen mixture under variable dosing

SUMMARY:
Low back pain is very common problem, variable modalities have been introduced to control such problem. One of the emerging modalities is the ozone - oxygen (O2-O3 ) mixture that could reduce the herniation disk size and inflammation.

DETAILED DESCRIPTION:
Intervertebral disc herniation is the most common problem which induces low back pain LBP. The number of patients seek surgical and or alternative therapy increases. The rate of re-operation is between 7-9% at 2 years and increases up to 10-25% at ten years postoperative.

Epidural injections with local anesthetics and steroids are one of the most commonly used interventions in managing chronic low back pain and lower extremity pain of various causes. However, despite their extensive use, debate continues on this medications effectiveness due to the lack of well-designed, randomized, controlled studies to determine the effectiveness of epidural injections in general, and caudal epidural injections in particular.

Ozone in mixture with oxygen has been justified in multiple studies have been done, this study aims to evaluate variable doses of this mix upon patient satisfaction, pain alleviation over 12 month follow up period .

ELIGIBILITY:
Inclusion Criteria:

* All patients Suffered radicular leg pain and some reported additional back pain.
* All patients are non-responsive to conservative treatment modalities with VAS more than 7.

Exclusion criteria

* presence of bleeding disorder
* local infection
* uncontrolled or degenerative spine disease
* pregnancy
* multilevel disk involvement
* patient refusal.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain alleviation by visual analogue scale (VAS) | 12 months
  assessing pain alleviation by visual analogue scale (VAS)

SECONDARY OUTCOMES:
Reduction of disk herniation by MRI | 6 months
  evaluation of disk herniation by MRI 6 month after injection, in comparison to the pre-injection MRI
Pain alleviation using Oswestry Low Back Pain Questionnaire | 12 months
  using Oswestry Low Back Pain Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elawamy A, Kamel EZ, Hassanien M, Wahba OM, Amin SE. Implication of Two Different Doses of Intradiscal Ozone-Oxygen Injection upon the Pain Alleviation in Patients with Low Back Pain: A Randomized, Single-Blind Study. Pain Physician. 2018 Jan;21(1):E25-E31. PMID 29357333